CLINICAL TRIAL: NCT07349056
Title: Evaluation of Periodontal Phenotype Following Orthognathic Surgery: A Two-Center, 6-Month Prospective Clinical and CBCT Study
Brief Title: Early Effects of Orthognathic Surgery on Periodontal Phenotype: A 6-Month Prospective Clinical and Radiographic Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: Trakya University (Other)
Collaborators: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Principal Investigator, Ece AÇIKGÖZ ALPARSLAN, Ass. Prof, Trakya University
Other Study IDs: 2522A04
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gingival Biotype; Gingival Phenotype; Buccal Bone Thickness; Recession, Gingival; Dental Surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Group A (Mandibular setback < 6 mm)
- Group B (Mandibular setback ≥ 6 mm)
- Group C (Mandibular advancement < 6 mm)
- Group D (Mandibular advancement ≥ 6 mm)
- Group E (Maxillary advancement < 6 mm + maxillary impaction)
- Group F (Maxillary advancement < 6 mm + maxillary downgrafting)
- Group G (Maxillary advancement < 6 mm + no impaction/downgrafting)
- Group H (Maxillary advancement ≥ 6 mm + maxillary impaction)
- Group I (Maxillary advancement ≥ 6 mm + maxillary downgrafting)
- Group J (Maxillary advancement ≥ 6 mm + no impaction/downgrafting)

SUMMARY:
The goal of this observational study is to learn how the health and thickness of the gums and supporting bone around the teeth change over 6 months in adults having jaw surgery to correct the bite. The main questions it aims to answer are:

* Do gum and tooth-support measurements change from before surgery to 1, 3, and 6 months after surgery?
* Do CT scan-based measurements of the tooth-supporting bone change over the same time period?

Participants will:

* Have a gum check-up (periodontal examination) before surgery and at 1, 3, and 6 months after surgery.
* Have CT scan-based measurements (CBCT) taken at the same time points for study assessment.

DETAILED DESCRIPTION:
This two-center prospective observational cohort study will enroll adult patients who are scheduled to undergo orthognathic surgery according to standard clinical indications. Orthognathic surgeries will be performed at Kocaeli Health and Technology University, while periodontal clinical examinations and CBCT-based assessments will be conducted at Trakya University. Participants will be evaluated at baseline (preoperatively) and at 1, 3, and 6 months after surgery. Clinical periodontal assessments will include predefined periodontal phenotype-related parameters recorded using a standardized protocol. CBCT datasets will be obtained and analyzed using a standardized measurement protocol to assess buccal alveolar bone-related parameters and the presence of dehiscence/fenestration where applicable. To minimize assessment bias, CBCT images will be coded and evaluated by an independent assessor blinded to surgical details and group classification, and clinical periodontal examinations will be performed by an examiner blinded to the surgical procedure details.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Presence of a Class III molar relationship of any severity at baseline.
* Presence of a Class II molar relationship of any severity at baseline.
* Presence of transverse arch discrepancies.
* Presence of vertical maxillary excess.
* Presence of maxillary and/or mandibular asymmetry.
* Presence of anterior open bite.
* Full permanent dentition up to the first molars, with no supernumerary teeth and no agenesis (congenital absence) of teeth up to the first molars.
* No previous orthodontic treatment.
* No history of tooth extraction other than second or third molars.
* Availability of complete baseline and end-of-follow-up periodontal parameters and phenotype records suitable for evaluation.
* Healthy periodontium with no signs of gingival hypertrophy.
* No systemic disease history or medication use that could affect gingival/periodontal conditions.

Exclusion Criteria:

* Patients planned for orthodontic camouflage treatment with fixed appliances for Class II/Class III correction instead of orthognathic surgery.
* History of interproximal enamel reduction (interproximal stripping).
* Presence of dental implants.
* Age < 18 years.
* Pregnant or breastfeeding individuals.
* Any systemic condition contraindicates orthognathic surgery.
* Psychiatric disorders.
* Syndromic conditions.
* History of previous orthognathic surgery.
* Refusal to sign the informed consent form.
* Individuals belonging to a vulnerable population.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred for orthognathic surgery to the Department of Oral and Maxillofacial Surgery at Kocaeli Health and Technology University and subsequently evaluated at the Department of Periodontology at Trakya University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-02-23 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
Change in width of keratinized gingiva (mm) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
  Width of keratinized gingiva is measured as the distance from the gingival margin to the mucogingival junction, recorded in mm.
Change in gingival thickness phenotype (thin vs thick) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
  Gingival thickness is assessed with a periodontal probe by the probe-transparency method and categorized as thin (≤1 mm; probe visible) or thick (>1 mm; probe not visible)
Change in buccal cortical bone thickness on CBCT (mm) | Baseline (preoperative) and postoperative follow-up CBCT records were obtained during routine controls (planned at 6 months).
  Buccal cortical bone thickness is measured on CBCT as the horizontal distance from the deepest point of the buccal marginal bone curvature (A) to the CEJ, and additionally at 4 mm apical to A and at the apex level, as defined in the protocol

SECONDARY OUTCOMES:
Probing pocket depth (mm) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
Bleeding on probing (0/1) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
Gingival Index (0-3) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
Plaque Index (0-3) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
Papilla loss classification (Nordland & Tarnow) | Baseline (preoperative) and postoperative 1, 3, and 6 months.
Gingival recession (mm) | Baseline and postoperative 1, 3, 6 months.
Fenestration/dehiscence presence on CBCT (yes/no) (and/or counts) | Baseline and postoperative 6 months.
Clinical attachment loss (mm) | Baseline and postoperative 1, 3, 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Trakya University Faculty of Dentistry, Edirne
  - Kocaeli Health and Technology University Faculty of Dentistry, Kocaeli

IPD SHARING:
Plan to Share IPD: No
Individual participant data containing personal health information will not be shared due to privacy and confidentiality requirements, as well as ethical restrictions and applicable standards